CLINICAL TRIAL: NCT06119958
Title: A Two-arm, Open-label, Single-sequence, Multiple Oral Dosings, Crossover Clinical Trial to Evaluate the Safety and the Pharmacokinetic Interaction of DWC202313 and DWC202314 in Healthy Adult Volunteers
Brief Title: Drug-drug Interactions Between DWC202313 and DWC202314 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DWJ1622101
Record Dates: First submitted 2023-10-23; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Drug Drug Interaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWC202313 (Experimental): DWC202313
  Interventions: Drug: DWC202313
- DWC202314 (Experimental): DWC202314
  Interventions: Drug: DWC202314

INTERVENTIONS:
Drug: DWC202313 — Experimental Drug 1
  Arms: DWC202313
Drug: DWC202314 — Experimental Drug 2
  Arms: DWC202314

SUMMARY:
This is A two-arm, open-label, single-sequence, multiple oral dosings, crossover study to evaluate the safety and the pharmacokinetic interaction of DWC202313 and DWC202314 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* over 19 year old

Exclusion Criteria:

* Galactose intolerance
* Lapp lactase deficiency

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Cmax,ss of DWC202313 and DWC202314 | Up to 14 days
AUCt,ss of DWC202313 and DWC202314 | Up to 14 days

SECONDARY OUTCOMES:
Tmax,ss of DWC202313 and DWC202314 | Up to 14 days
Cmin,ss of DWC202313 and DWC202314 | Up to 14 days
t1/2 of DWC202313 and DWC202314 | Up to 14 days
CLss/F of DWC202313 and DWC202314 | Up to 14 days
Vdss/F of DWC202313 and DWC202314 | Up to 14 days
PTF of DWC202313 and DWC202314 | Up to 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus YANGJI Hospital, Seoul, South Korea